CLINICAL TRIAL: NCT00593138
Title: A Randomized Open-label Study of Dopamine Transporter Receptor Occupancy With Long-acting Dex-methylphenidate (20 mg, 30 mg, and 40 mg) as Measured With C-11 Altropane in Healthy Adult Volunteers
Brief Title: Study of Dopamine Transporter Receptor Occupancy With Long-acting Dex-methylphenidate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Associate Chief, Clinical and Research Program, Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2006-p-001610
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Drug Binding to DAT Receptors
Keywords: Focalin XR; Adult; PET scan
MeSH Terms: interventions — Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: dex-methylphenidate

INTERVENTIONS:
Drug: dex-methylphenidate — The drug is administered as a capsule by mouth. Participants are assigned to receive either 20, 30 or 40 mg doses before each scan visit.
  Other Names: Focalin XR

SUMMARY:
The objectives of this study are to document the pharmacokinetics of the adequacy of DAT receptor occupancy d-MPH formulation in three doses (20 mg, 30 mg, and 40 mg) using PET scanning with C-11 Altropane as the ligand across a range of times. It has been estimated that MPH is effective when the average CNS DAT occupancy is 50% or greater. Focalin XR has been shown to be clinically effective in an analog classroom as early as 1 hour and as late as 12 hours. Therefore, it is hypothesized that the average DAT occupancy will be adequate (50% or greater) at time periods corresponding to the times of clinical efficacy.

The first objective is to examine the onset of action by testing whether average DAT occupancy will be adequate (50% or greater) at 1 hour after dosing for each dose tested (20 mg, 30 mg, 40 mg).

The second objective is to test the adequacy of average DAT occupancy in a range of later times for each dose. The times chosen (8, 10 and 12 hours) correspond to times Focalin XR has been shown to be clinically effective in an analogue classroom study. A range of times have been chosen since, while effective at 12 hours, the degree of clinical effectiveness decreased with later time periods. The adequacy of DAT occupancy across this range of time periods will provide important details on the in vivo molecular action of the medicine at periods of critical clinical activity.

The third exploratory objective is to examine a time period later then those previously tested with the highest dose. Since the clinical effectiveness of Focalin XR has not been tested out to 14 hours, it is unknown whether it is effective at 14 hours. If Focalin XR were to be effective at 14 hours it would be more likely at the highest dose.

DETAILED DESCRIPTION:
Stimulants have been shown to be very effective in the treatment of Attention Deficit Hyperactivity Disorder (ADHD). [1] Studies have shown that full day treatment is often preferable to shorter treatment [2] and recent guidelines advise full day treatment. [3] However, there are many barriers to giving multiple doses of short acting medicine. New delivery systems have evolved to overcome tachyphylaxis and provide effective long-acting treatment with a single pill. [4] One of the new formulations is the spheroidal oral drug absorption system (SODAS). SODAS consists of capsules with two types of beads in a 1 to 1 ratio. One type of bead provides immediate release methylphenidate (IR MPH), and the other type of bead consists of MPH coated with a polymer that delays release for 4 hours. SODAS MPH has been shown to be effective in clinical studies [5]. However, the mechanism of action remains unclear. While pharmacokinetic studies have shown a double pulse profile in the serum [4], the central nervous system pharmacokinetics are unknown. Understanding the central nervous system pharmacokinetic properties is critical for new drug development for ADHD, especially for drugs of different lengths of action.

The d-MPH form has been shown to be the active enantiomer of MPH. Studies have shown that the duration of action of d-MPH is longer than that of racemic MPH. Clinical studies of once a day d-MPH has demonstrated efficacy in children, adolescents and adults with ADHD. Understanding the central nervous system pharmacokinetic properties of the SODAS formulation of the longer-acting (d) enantiomer will provide critical knowledge of its mechanism of action.

The main target of MPH in the brain is the dopamine transporter (DAT) [6]. There is now an exquisitely sensitive methodology to measure DAT occupancy using C-11 Altropane and Positron Emission Tomography (PET) [7]. The time course of decay of the C-11 Altropane permits repeated imaging, thus allowing documentation of the pharmacokinetics of DAT receptor occupancy. A group at Massachusetts General Hospital has previously documented the central nervous system pharmacokinetics of several psychiatric drugs using similar techniques [8-12].

To this end, this protocol seeks to document the pharmacokinetics of DAT receptor occupancy of d-MPH using PET and C-11 Altropane. It has been estimated that MPH is effective when the CNS DAT occupancy is 50% or greater. This aim of this study will be to measure CNS DAT occupancies at extended time points after administration of d-MPH. This research will provide novel and unique information toward a better understanding of the mechanism of action of long-acting stimulant formulations to enable new drug development.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to participate in the study.
2. Age: 18 -45, inclusive
3. If female, non-pregnant, non-nursing with a negative serum pregnancy test.
4. Female subjects will agree to use an acceptable and effective form of birth control during the course of their study participation.
5. Supine and standing blood pressure < 150/90 mmHg.
6. Heart rate, after resting for 5 minutes, within the range 46-90 beats/min.
7. Right handed.

Exclusion Criteria:

1. Diagnosis of any psychotic disorder, bipolar disorder, severe depression, severe anxiety, or Autism. Subjects with mild mood, oppositional, conduct, and anxiety disorders may be permitted to participate if considered appropriate by the investigator.
2. Scores of Baseline Scales:

   * Hamilton Depression Scale > 12 (out of a possible 67 on the 21-item scale)[18]
   * Beck Depression Inventory > 19 (out of a possible 63 on the 21-item scale)[19]
   * Hamilton Anxiety Scale > 21 (out of a possible 56 on the 14-item scale) [20]
3. Subjects with motor tics or with a family history or diagnosis of Tourette's Syndrome.
4. History of head trauma with loss of consciousness, organic brain disorders, seizures, or neurosurgical intervention.
5. Any clinically significant chronic medical condition, in the judgment of the investigator.
6. In the judgment of the investigator, has a mental impairment as evidenced by an I.Q. <75.
7. Exposure to dopamine receptor antagonists within the previous three (3) months.
8. Exposure to radiopharmaceuticals within four (4) weeks prior to PET scan.
9. Subjects receiving psychotropic medication including MAO inhibitors within the past 6 to 12 months.
10. Any clinically significant abnormality in the screening laboratory tests, vital signs, or 12 lead ECG, outside of normal limits.
11. Any pre-existing structural cardiac abnormalities.
12. A history or known family history of long QT syndrome or QTc >450 ms (males) or >470 ms (females).
13. Any family history of cardiac sudden death.
14. QTc prolongation of QTc > 450 ms (male) or 470 ms (female), hypertension or cardiac arrhythmia, or increased heart rate for age in the judgment of the investigator at screening.
15. A history of cardiac structural abnormality
16. Any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant.
17. Subjects with a known recent history (within the past six (6) months) of illicit drug or alcohol dependence.
18. Subjects diagnosed with glaucoma.
19. Subjects at risk for MPH toxicity (e.g. individuals with arrhythmias, coronary artery disease, etc.).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
DAT occupancy from PET scan results | each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Spencer TJ, Bonab AA, Dougherty DD, Mirto T, Martin J, Clarke A, Fischman AJ. Understanding the central pharmacokinetics of spheroidal oral drug absorption system (SODAS) dexmethylphenidate: a positron emission tomography study of dopamine transporter receptor occupancy measured with C-11 altropane. J Clin Psychiatry. 2012 Mar;73(3):346-52. doi: 10.4088/JCP.10m06393. Epub 2011 Nov 1. PMID 22154896